CLINICAL TRIAL: NCT04302025
Title: NAUTIKA1: A Multicenter, Phase II, Neoadjuvant and Adjuvant Study of Multiple Therapies in Biomarker-selected Patients With Resectable Stages IB-III Non-small Cell Lung Cancer
Brief Title: A Study of Multiple Therapies in Biomarker-selected Participants With Resectable Stages IB-III Non-small Cell Lung Cancer (NSCLC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML41591
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — alectinib; entrectinib; Vemurafenib; cobimetinib; pralsetinib; atezolizumab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- ALK Cohort (Enrolment Closed) (Experimental): Participants will receive up to 8 weeks of alectinib neoadjuvant treatment before undergoing surgical resection per standard of care (SOC). All participants that undergo surgical resection and whose tumors have pathological response or lack radiographic progression will be eligible for the adjuvant treatment phase with alectinib. Adjuvant therapy will consist of 4 cycles of chemotherapy followed by up to 2 years of alectinib.
  Enrolment Closed.
  Interventions: Drug: Alectinib; Procedure: Resection; Drug: Chemotherapy
- ROS 1 Cohort (Enrolment Closed) (Experimental): Participants will receive up to 8 weeks of entrectinib neoadjuvant treatment before undergoing surgical resection per SOC. All participants that undergo surgical resection and whose tumors have pathological response or lack radiographic progression will be eligible for the adjuvant treatment phase with entrectinib. Adjuvant therapy will consist of 4 cycles of chemotherapy followed by up to 2 years of entrectinib.
  Enrolment Closed.
  Interventions: Drug: Entrectinib; Procedure: Resection; Drug: Chemotherapy
- NTRK Cohort (Enrolment Closed) (Experimental): Participants will receive up to 8 weeks of entrectinib neoadjuvant treatment before undergoing surgical resection per SOC. All participants that undergo surgical resection and whose tumors have pathological response or lack radiographic progression will be eligible for the adjuvant treatment phase with entrectinib. Adjuvant therapy will consist of 4 cycles of chemotherapy followed by up to 2 years of entrectinib.
  Enrolment Closed.
  Interventions: Drug: Entrectinib; Procedure: Resection; Drug: Chemotherapy
- BRAF Cohort (No Participants Enrolled, Cohort Closed) (Experimental): Participants will receive up to 8 weeks of vemurafenib plus cobimetinib neoadjuvant treatment before undergoing surgical resection per SOC. All participants that undergo surgical resection and whose tumors have pathological response or lack radiographic progression will be eligible for the adjuvant treatment phase with vemurafenib plus cobimetinib. Adjuvant therapy will consist of 4 cycles of chemotherapy followed by up to 2 years of of vemurafenib plus cobimetinib.
  Cohort closed.
  Interventions: Drug: Vemurafenib; Drug: Cobimetinib; Procedure: Resection; Drug: Chemotherapy
- RET Cohort (Cohort closed) (Experimental): Participants will receive up to 8 weeks of pralsetinib neoadjuvant treatment before undergoing surgical resection per SOC. All participants that undergo surgical resection and whose tumors have pathological response or lack radiographic progression will be eligible for the adjuvant treatment phase with pralsetinib. Adjuvant therapy will consist of 4 cycles of chemotherapy followed by up to 2 years of pralsetinib.
  Cohort closed.
  Interventions: Drug: Pralsetinib; Procedure: Resection; Drug: Chemotherapy
- PD-L1 Cohort (Enrolment Closed) (Experimental): Participants with positive programmed death-ligand 1 (PD-L1) in ≥1% tumor cells will receive 4 cycles of atezolizumab neoadjuvant treatment. During neoadjuvant Cycle 1 of atezolizumab, participants will also receive low-dose stereotactic body radiation therapy (SBRT) (8 gray [Gy] X 3). Adjuvant treatment consists of SOC treatment as determined by the investigator, per National Comprehensive Cancer Network (NCCN) guidelines.
  Enrolment Closed.
  Interventions: Drug: Atezolizumab; Drug: SBRT; Procedure: Resection
- KRAS G12C Cohort (Experimental): Participants will receive up to 8 weeks of divarasib as neoadjuvant treatment before undergoing surgical resection per SOC. PD-L1 negative participants whose tumors have pathological response or lack radiographic progression will be have the option of continuing divarasib alone for up to 3 years or 1-4 cycles of SOC chemotherapy followed by divarasib for 3 years as adjuvant therapy. For participants who test positive PD-L1, they will have the option to receive 1-4 cycles of SOC chemotherapy followed by atezolizumab for up to 16 cycles or SOC alone.
  Interventions: Procedure: Resection; Drug: Chemotherapy; Drug: Divarasib

INTERVENTIONS:
Drug: Alectinib — Participants will receive oral alectinib twice per day (BID).
  Arms: ALK Cohort (Enrolment Closed)
Drug: Entrectinib — Participants will receive oral entrectinib daily.
  Arms: NTRK Cohort (Enrolment Closed); ROS 1 Cohort (Enrolment Closed)
Drug: Vemurafenib — Participants will receive oral vemurafenib BID.
  Arms: BRAF Cohort (No Participants Enrolled, Cohort Closed)
Drug: Cobimetinib — Participants will receive oral cobimetinib daily.
  Arms: BRAF Cohort (No Participants Enrolled, Cohort Closed)
Drug: Pralsetinib — Participants will receive oral pralsetinib daily.
  Arms: RET Cohort (Cohort closed)
Drug: Atezolizumab — Atezolizumab will be administered by intravenous (IV) infusion.
  Arms: PD-L1 Cohort (Enrolment Closed)
Drug: SBRT — Participants will receive SBRT given concurrently, starting with the first dose of atezolizumab.
  Arms: PD-L1 Cohort (Enrolment Closed)
Procedure: Resection — Participants will receive surgical resection of the primary tumor along with selected lymph nodes per SOC.
Drug: Chemotherapy — Participants will receive SOC chemotherapy as determined by the treating physician.
  Arms: ALK Cohort (Enrolment Closed); BRAF Cohort (No Participants Enrolled, Cohort Closed); KRAS G12C Cohort; NTRK Cohort (Enrolment Closed); RET Cohort (Cohort closed); ROS 1 Cohort (Enrolment Closed)
Drug: Divarasib — Participants in the KRAS G12C cohort will receive oral divarasib for approximately 8 weeks until the day before surgery as neoadjuvant therapy up to 3 years as adjuvant therapy.
  Arms: KRAS G12C Cohort

SUMMARY:
This trial will evaluate the efficacy and safety of various therapies in participants with Stage IB, IIA, IIB, IIIA, or selected IIIB resectable and untreated NSCLC tumors that meet protocol-specified biomarker criteria.

ELIGIBILITY:
Inclusion Criteria for Neoadjuvant Therapy:

* Pathologically documented NSCLC:
* Newly diagnosed early-stage NSCLC stages IB, IIA, IIB, IIIA, or selected IIIB (T3N2 only) NSCLC of squamous or non-squamous histology. Staging should be based on the 8th edition of the American Joint Committee on Cancer (AJCC)/Union Internationale Contre le Cancer (UICC) NSCLC staging system
* T4 primary NSCLC will be allowed only on the basis of size. Invasion of the diaphragm, mediastinum, heart, great vessels, trachea, recurrent laryngeal nerve, esophagus, vertebral body, carina, and separate tumor nodules in a different ipsilateral lobe is not permitted
* All participants will undergo clinical staging using computed tomography (CT) and positron emission tomography (PET) scanning, as well as brain imaging using magnetic resonance imaging (MRI). Invasive mediastinal staging by either mediastinoscopyor endo- bronchial ultrasonography is highly encouraged for participants with radiographically suspected mediastinal nodal disease (ie, N2) but not mandated if the CT or PET scans showed no evidence of N2 disease
* Molecular testing results from clinical laboratory improvement amendments (CLIA)-certified laboratories and showing at least one of the following abnormalities: ALK fusion, ROS1 fusion, NTRK1/2/3 fusion; BRAF V600 mutation, RET fusion, PD-L1 expression in ≥ 1% tumor cells as determined by FDA-approved test, KRAS G12C mutation
* Measurable disease, as defined by RECIST v1.1
* NSCLC must have a solid or subsolid appearance on CT scan and cannot have a purely ground glass opacity appearance. For subsolid lesions, the tumor size (i.e., clinical T stage) should be measured based on the solid component only, exclusive of the ground glass opacity component
* Evaluated by the attending surgeon prior to study enrollment to verify that the primary tumor and any involved lymph nodes are technically completely resectable and verify that the participant is medically operable
* Adequate pulmonary function to be eligible for surgical resection with curative intent
* Adequate cardiac function to be eligible for surgical resection with curative intent
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Adequate hematologic and end-organ function
* Negative hepatitis B surface antigen (HBsAg) test at screening for cohort
* Negative total hepatitits B core antibody (HBcAb) test at screening for cohort, or positive total HBcAb test followed by a negative hepatitis B virus (HBV) deoxyribonucleic acid (DNA) test at screening
* Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV ribonucleic acid (RNA) test at screening
* Male participants must be willing to use acceptable methods of contraception
* Female participants of childbearing potential must agree to use acceptable methods of contraception

Inclusion Criteria for Adjuvant Therapy (TKI Cohorts and KRAS G12C cohort [if continuing on Divarasib]):

* Participants whose tumors lack radiographic progression
* ECOG Performance Status of 0 or 1
* Adequate hematologic and end-organ function

Exclusion Criteria

* NSCLC that is clinically T4 by virtue of mediastinal organ invasion or Stage IIIB by virtue of N3 disease
* Any prior therapy for lung cancer, including chemotherapy, targeted therapy, immunotherapy, or radiotherapy, within 2 years
* Participants with prior lung cancer
* Major surgical procedure within 28 days prior to Cycle 1, Day 1
* Malignancies other than the disease under study within 3 years prior to Cycle 1, Day 1, with the exception of participants with a negligible risk of metastasis or death and with expected curative outcome
* Treatment with an investigational agent for any condition within 4 weeks prior to Cycle 1, Day 1
* Participants known to be positive for human immunodeficiency virus (HIV) are excluded if they meet any of the following criteria: cluster of differentiation 4 (CD4)+ T-cell count of <350 cells/microliters (cells/µL); detectable HIV viral load; history of an opportunistic infection within the past 12 months; on stable antiretroviral therapy for <4 weeks
* Severe infection within 4 weeks prior to initiation of study treatment, including but not limited to hospitalization for complications of infections, or any active infection that, in the opinion of the investigator, could impact participant safety
* Pregnant or lactating, or intending to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2020-11-06 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2030-05-30 (Estimated)

PRIMARY OUTCOMES:
Tyrosine Kinase Inhibitor (TKI) Cohort: Proportion of Participants With Major Pathologic Response (MPR) | After surgical resection (approximately study Week 8)
  MPR is defined as ≤ 10% residual viable tumor cells as scored by local pathologists.
Checkpoint Inhibitor (CPI) Cohort: Pathological Complete Response (pCR) | After surgical resection (approximately study Week 8)
  Scored by local pathologists; defined as lack of any viable tumor cells on review of hematoxylin and eosin (H&E) slides after complete evaluation of a resected lung cancer specimen including all sampled regional lymph nodes.
KRAS Cohort: Percentage of Participants With 3-5 Grade Adverse Events (AEs) | After surgical resection (approximately study Week 8)
KRAS Cohort: Percentage of Participants Without Delays of Surgery due to Treatment-related Adverse Events as Reported by the Investigator | After surgical resection (approximately study Week 8)

SECONDARY OUTCOMES:
Proportion of Participants With MPR | After surgical resection (approximately study Week 8)
  Defined as ≤10% residual viable tumor cells) based on surgical resection as defined by Hellmann et al. (2014) and Travis et al. (2020). TKI cohorts: MPR will be scored by a central pathology committee consensus read. CPI cohort: MPR will be scored by local pathologists and central pathology committee consensus read. KRAS G12C cohort: MPR will be scored by local pathologists and central pathology committee consensus read.
Proportion of Participants With pCR | After surgical resection (approximately study Week 8)
  Defined as lack of any viable tumor cells on review of H&E slides after complete evaluation of a resected lung cancer specimen, including all sampled regional lymph nodes.
  TKI cohorts: pCR will be scored by local pathologists and a central pathology committee consensus read.
  CPI cohort: pCR will be scored by a central pathology committee consensus read. KRAS G12C cohort: pCR will be scored by a central pathology committee consensus read.
Pathological Regression Based on Weighted % Viable Tumor Cell Assessment | After surgical resection (approximately study Week 8)
Investigator-assessed Response Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | After neoadjuvant treatment (after approximately study Week 8)
Pathological Complete Response (pCR) as Assessed by Local and Central Pathology Laboratories | At the time of surgical resection (approximately study Week 8)
  Defined as the absence of any viable tumor in main tumor bed at the time of surgical resection, as assessed by local and central pathology laboratories.
Disease-free Survival (DFS) | From the first date of no disease to local or distant recurrence or death from any cause, whichever occurs first, through the end of the study (up to 9 years)
Event-free Survival (EFS) | From first dose of study treatment to first documented disease progression per RECIST v1.1, or local or distant disease recurrence as determined by investigator, or death from any cause, whichever occurs first, through the end of study (up to 9 years)
Overall Survival (OS) | From the first dose of study medication to death from any cause, through the end of the study (up to 9 years)
Percentage of Participants With Adverse Events (AEs) | Up to 9 years
Nodal Downstaging | After surgical resection (approximately study Week 8)
  Defined as percentage of participants with reduced stages in regional lymph nodes at surgery.
Circulating tumor DNA (ctDNA) Clearance Rate | Prior to surgery (before study Week 8)
KRAS G12C Cohort: Plasma Concentration of Divarasib at Specified Timepoints | Cycle 1 Day 1, Cycle 2 Day 1 (Cycle= 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (38):
- United States (38):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope - Orange County Lennar Foundation Cancer Center, Irvine, California
  - USC Norris Cancer Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Los Angeles - Jonsson Comprehensive Cancer Center, Los Angeles, California
  - The Center for Cancer Prevention and Treatment at St.Joseph Hospital of Orange, Orange, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Helen Diller Family CCC, San Francisco, California
  - University of Colorado - Anschutz Medical Campus (University of Colorado Health Sciences Center), Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - MedStar Georgetown University Hospital (Lombardi Comprehensive Cancer Center), Washington D.C., District of Columbia
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Boston Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute - Farmington Hills/Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center - Washington University Medical Campus, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Laura and ISAAC Perlmutter Cancer Center at NYU Langone., New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - AHN Cancer Institute ? Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Baptist Clinical Research Institute, Memphis, Tennessee
  - Tennessee Oncology - Nashville, Nashville, Tennessee
  - Kelsey Seybold Clnic, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Lumi Research, Kingwood, Texas
  - Virginia Cancer Specialists (Fairfax) - USOR, Fairfax, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing